CLINICAL TRIAL: NCT03893461
Title: Impact of Stereotactic Body Radiation Therapy on the Coagulation System in Patients With Non-small Cell Lung Cancer
Brief Title: Coagulation System In STereotactic Radiotherapy Of NSCLC
Acronym: CISTRON
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Stefan Starup Jeppesen, MD, PhD, Odense University Hospital
Other Study IDs: S-20180109
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Thromboembolism; Lung Cancer; NSCLC; Radiotherapy; Complications
MeSH Terms: conditions — Thromboembolism; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample collection for biobank
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: x — Stereotactic body radiation therapy for localized NSCLC

SUMMARY:
The risk of thromboembolism is elevated in lung cancer patients. The present project investigates whether stereotactic body radiation therapy (SBRT) further increases the risk of thromboembolic disease in lung cancer patients.

If coagulation is activated by SBRT, this study could form the basis of new clinical trials investigating whether lung cancer patients may benefit from thromboprophylaxis during and after stereotactic body radiation therapy.

DETAILED DESCRIPTION:
In this study, the patients will have blood samples drawn three times (prior to start of stereotactic body radiation therapy, immediately after stereotactic body radiation therapy completion, four to six weeks after completing stereotactic body radiation therapy). The blood sample at the completion of stereotactic body radiation therapy is an extra compared to normal gathering of blood samples of patients with NSCLC treated with stereotactic body radiation therapy. Also extra glasses with blood will be gathered at each blood sample for storage in a biobank in order to be able to make future analysis on this material.

There is a minimal risk of developing infection or hematoma in connection with blood sampling but we consider this risk to be negligible. The total volume of 120 ml blood drawn over a period of 6 weeks is an inconsiderable risk for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Planned stereotactic body radiation therapy of lung cancer

Exclusion Criteria:

* Inability to provide informed consent
* Venous thrombosis within the last three months
* Active cancer within the previous year except for lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective study of 100 consecutively included lung cancer patients receiving stereotactic body radiation therapy. As standard treatment, which is considered for best practice, the patients receive:
  1. 66 Gy/ 3 fractions (F) (new primary peripheral lung cancer), or
  2. 50 Gy/ 5 F (new primary central lung cancer), or
  3. 45 Gy/ 3 F (peripheral lung cancer relapse after initial surgery or stereotactic body radiation therapy)
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in coagulation | From start of SBRT to end and 5 weeks after SBRT
  endogenous thrombin

CONTACTS AND LOCATIONS:
Overall Officials: Stefan S Jeppesen, MD, PhD, Principal Investigator — Department of Oncology, Odense University Hospital
Locations (1):
- Department of Oncology, Odense University Hospital, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: Undecided